CLINICAL TRIAL: NCT02557087
Title: Efficacy of Intravenous Hyoscine ButylBromide as an Analgesic During the First Stage of Labor: A Randomized Controlled Trial
Brief Title: Hyoscine ButylBromide for Intrapartum Analgesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Bakry Mohye Soliman El Kinawy, TA, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP-HBB
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Analgesia, Obstetrical
MeSH Terms: conditions — Agnosia | interventions — Scopolamine; Meperidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyoscine (Experimental): Intravenous administration of Hyoscine N-butylbromide diluted in 10 mL of sterile water (single dose), as an analgesic during the first stage of labor, given by a member of the study team.
  Interventions: Drug: Hyoscine
- Pethidine (Active Comparator): Slow intravenous administration of pethidine, 50 mg to be diluted in 10 mL of sterile water (single dose), as an analgesic during the first stage of labor, given by a member of the study team.
  Interventions: Drug: Pethidine

INTERVENTIONS:
Drug: Hyoscine
  Arms: Hyoscine
Drug: Pethidine
  Arms: Pethidine

SUMMARY:
The aim of this study is to assess whether hyoscine butylbromide is as effective as pethidine for analgesia during the first stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Primiparity
* Active phase of labor (cervical dilatation of 3-5 cm, in the presence of adequate uterine contractions; lasting at least 40 seconds at intervals of 3-4 minutes)
* Maternal age between 20-30 years
* Singleton term pregnancy (37-42 weeks of gestation)
* Vertex-presenting fetus

Exclusion Criteria:

* Clinical evidence of cephalopelvic disproportion.
* Scarred uterus; previous cesarean section, hysterotomy or myomectomy.
* Any medical disorders associated with pregnancy.
* Fetal distress
* Receiving any regional or parenteral analgesia before recruitment in the study
* Known hypersensitivity to the drug family

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The efficacy of intravenous tenoxicam to supply adequate analgesia as indicated by changes in the pain intensity score using the visual analog scale. | 4 hours
  Assessment is to be done and followed up by the investigator at ½, 1, 2, 3 and 4 hours from drug administration. Scores range from 0 [no pain] to 10 [worst possible pain].